CLINICAL TRIAL: NCT02299687
Title: A Clinical Trial to Investigate the Influence of CYP2C19 Polymorphism on Pharmacokinetic/Pharmacodynamic Characteristics of Omeprazole in Healthy Korean Volunteers
Brief Title: Influence of CYP2C19 Polymorphism on PK/PD of Omeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In-Jin Jang, MD, PhD, Professor of clinical pharmacology, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OMP_CYP2C19
Record Dates: First submitted 2014-09-21; First posted 2014-11-24 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Stomach Ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — Omeprazole

ARMS (3):
- CYP2C19 EM (Experimental): CYP2C19 EM
  Interventions: Drug: Omeprazole
- CYP2C19 IM (Experimental): CYP2C19 IM
  Interventions: Drug: Omeprazole
- CYP2C19 PM (Experimental): CYP2C19 PM
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole

SUMMARY:
A clinical trial to investigate the influence of CYP2C19 polymorphism on pharmacokinetic/pharmacodynamic characteristics of omeprazole in healthy Korean volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Are able to provide written informed consent.
2. The subject is a healthy Korean aged 20 to 45 years, inclusive.
3. The subject weighs at least 55 (for female, 55) to 90 kg and has a body mass index (BMI) range of 18 to 25 kg/m2

Exclusion Criteria:

1. Subjects with evidence or a history of clinically significant pulmonary, cardiovascular, hepatic, endocrine, hematological, neurologic or psychiatric diseases.
2. Subjects with evidence of gastrointestinal disease which can affect the absorption of drug.
3. Subjects with a history of drug abuse or a positive result in the urine drug screening for drug abuse
4. Subjects who have taken any prescribed medicine or herbal medicine within 2 weeks before the first administration of the investigational product, any non-prescribed medicine or vitamin supplement within 1 week prior the first administration of the investigational product (if all other conditions are satisfied, subjects may be eligible for the trial as judged by the investigator.)
5. Subjects who have donated a unit of whole blood within 30 days or who have participated in any other clinical trial within 60 days prior the first administration of the investigational product
6. Subject who have history of allergy on omeprazole
7. Subject who can not continue proper contraception method during study period.
8. Subject with a positive urine HCG test result on screening. (in case of woman subject)
9. Subjects who consume more than 21 units of alcohol per week (1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking during the PK/PD testing period
10. Subjects who consume more than 10 cigarette per day or who are unable to abstain from smoking during the PK/PD testing period
11. Subjects who are unable to abstain from grapefruit or caffeine containing food 3 day prior the first administration of the investigational product
12. Subjects judged not eligible for the study after reviewing the clinical laboratory results or other reasons by the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
mean and median Intragastric PH | 24 hour

SECONDARY OUTCOMES:
AUC | 12 hour
Cmax | 12 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park S, Hyun YJ, Kim YR, Lee JH, Ryu S, Kim JM, Oh WY, Na HS, Lee JG, Seo DW, Hwang IY, Park Z, Jang IJ, Oh J, Choi SE. Effects of CYP2C19 Genetic Polymorphisms on PK/PD Responses of Omeprazole in Korean Healthy Volunteers. J Korean Med Sci. 2017 May;32(5):729-736. doi: 10.3346/jkms.2017.32.5.729. PMID 28378544